CLINICAL TRIAL: NCT06110858
Title: The Efficacy of Tinkering Activity Based Cognitive Intervention to Improve Executive Function in Individuals With Subjective Cognitive Decline：A Pilot Study
Brief Title: Efficacy of Tinkering Activities in Individuals With Subjective Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan Science Education Center(NTSEC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202310004RIND
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Training; Subjective Cognitive Decline
Keywords: Subjective Cognitive Decline; Cognitive Intervention; Executive Function; Problem Solving; Cognitive Flexibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tinkering Activities (Experimental)
  Interventions: Behavioral: Tinkering Activities

INTERVENTIONS:
Behavioral: Tinkering Activities — Tinkering activities encompass elements of science, art and technology. They emphasize that learning is not simply about teachers imparting knowledge to students, but rather about students actively constructing knowledge themselves. Tinkering activities are characterized by three key elements: active engagement, open-ended exploration and problem-solving. In such activities, participants are provided with products without telling the steps. They are then encouraged to attempt creating it on their own. During this hands-on learning process, participants need to flexibly change their mindset, think outside the box and tackle emerging problems, which challenge their executive functions.

SUMMARY:
Given that preventing and delaying the onset of dementia is a crucial public health policy issues worldwide, it is essential to develop effective interventions and implement early interventions before the onset of dementia. Subjective Cognitive Decline (SCD) is considered the earliest manifestation of dementia and individuals with SCD may have a higher risk for future cognitive decline and dementia. Despite performing normally on objective cognitive tests, individuals with SCD have been found to exhibit worse performance on some cognitive domains, including executive functions, compared to those without SCD. Executive Functions (EFs) refer to a set of cognitive processes that include working memory, inhibition, cognitive flexibility, planning, problem solving and reasoning, enabling individuals to achieve goals by controlling and regulating thoughts and behaviors. EFs are important for our daily functioning and their decline can negatively impact an individual's quality of life. However, to our knowledge, there is limited research on maintaining or improving EFs in individuals with SCD. Tinkering Activity (TA) is a hands-on cognitive activity that emphasizes process of problem-solving, active engagement and open-ended exploration, which challenges EFs. In addition, previous research has shown the benefits of TA for community-dwelling older adults.

Therefore, the goal of this clinical tri is to examine the efficacy of TA based cognitive intervention in enhancing EFs in individuals with SCD. This study will be a one-group pretest-posttest design. Twelve to fifteen individuals with SCD will be recruited from the communities. All participants will receive 12 intervention sessions, each lasting 2 hours, with two sessions per week for 6 weeks. All participants will be assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years
* Can communicate in Mandarin and is literate in Chinese
* No impairment in basic activities of daily living(BADL) or Barthel Index score of 100
* Score >23 on the Taiwanese version of the Montreal Cognitive Assessment(MoCA-T)
* Willing and able to participate fully in the intervention
* Individuals with Subjective Cognitive Decline, screened from the communities:

  1. Experience subjective cognitive difficulties: answered "yes" to any questions in part I of the Subjective Cognitive Decline Scale(SCDS).
  2. Display normal performance in the Color Trails Test and Word Lists Test of the Wechsler Memory Scale-3rd Edition(after adjustment of age, gender and education, scoring on average above -1.5 standard deviations)

Exclusion Criteria:

* Diagnosed with Mild Cognitive Impairment(MCI) or Dementia
* Cognitive changes due to psychiatric or neurological disorders, substance abuse, and those with unstable conditions and symptomatic disturbances, or a score of ≥ 29 on the Beck Depression Inventory II (BDI-II)
* Unable to participate due to physical illnesses
* Severe impairment in visual and auditory abilities
* Participated in other cognitive training while engaged in this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Changes of Tower of Hanoi task(TOH) | Week 0, Week 6
  Scoring takes into account the number of movements, completion times, and the number of violations. Fewer movements, shorter completion times, and fewer violations indicate better planning and problem-solving.
Changes of Task Switching Paradigm(TS) | Week 0, Week 6
  Scoring takes into account reaction time and accuracy. Faster reaction times and higher accuracy indicate better cognitive flexibility.
Changes of Colour Trails Test-2(CTT-2) | Week 0, Week 6
  Scoring takes into account times, colour errors, number errors, near-misses and prompts. Fewer times, colours errors, number errors, near-misses and prompts indicate better cognitive flexibility.

SECONDARY OUTCOMES:
Changes of Guilford's Alternative Uses Task(GAU) | Week 0, Week 6
  Scoring includes criteria such as originality, fluency, flexibility and elaboration. A higher score indicates better creativity and divergent thinking.
Changes of Remote Associates Test(RAT) | Week 0, Week 6
  Scoring ranges from 0 to 30. A higher score indicates better remote associate ability.
Changes of the Brief University of California San Diego Performance-Based Skills Assessment-Traditional Chinese Version(UPSA-B) | Week 0, Week 6
  Scoring ranges from 0 to100. A higher score indicates better performance in instrumental activities of daily living.
Changes of Computerized Everyday Cognitive Function Assessment(CECFA) | Week 0, Week 6
  Scoring takes into account both correct rate and time. A higher score indicates better performance in instrumental activities of daily living.
Changes of the Taiwanese version of the Montreal Cognitive Assessment(MoCA-T) | Week 0, Week 6
  Scoring ranges from 0 to 30. A higher score indicates better objective cognitive function.
Changes of Subjective Cognitive Decline Scale(SCDS) | Week 0, Week 6
  Scoring ranges from 14 to 70. A higher score indicates individuals perceive more subjective cognitive difficulties.
Changes of Word Lists Test(WLT) in Wechsler Memory Scale-3rd Edition(WMS-III) | Week 0, Week 6
  Scoring includes part I(WLT-I) and part II(WLT-II). WLT-II is administered 25-35 minutes after WLT-I. A higher score indicates better verbal short term and long-term memory.
Changes of Family Pictures(FP) in Wechsler Memory Scale-3rd Edition(WMS-III) | Week 0, Week 6
  Scoring includes part I(FP-I) and part II(FP-II). FP-II is administered 25-35 minutes after WLT-I. A higher score indicates better visual short term and long-term memory.
Changes of Colour Trails Test-1(CTT-1) | Week 0, Week 6
  Scoring takes into account times, errors, near-misses and prompts. Fewer times, errors, near-misses and prompts indicate better attention.
Changes of Beck Depression Inventory II(BDI-II) | Week 0, Week 6
  Scoring ranges from 0 to 63. A higher score indicates individuals perceive more severe depressive symptoms.
Changes of Beck Anxiety Inventory(BAI) | Week 0, Week 6
  Scoring ranges from 0 to 63. A higher score indicates individuals perceive more severe anxiety symptoms.
Changes of General Self-Efficacy Scale(GSE) | Week 0, Week 6
  Scoring ranges from 10 to 40. A higher score indicates better self-efficacy.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University, Taipei
  - School of Occupational Therapy, College of Medicine, National Taiwan University, Taipei

IPD SHARING:
Plan to Share IPD: No